CLINICAL TRIAL: NCT05175391
Title: Improving the Liking and Consumption of Protein Rich Foods in Older Adults Through the Use of Culinary Spices
Brief Title: Improving Protein Intake in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 21-3652
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Food Preferences
Keywords: taste test; spices; food liking; protein
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: To determine the consumption, liking, flavor intensity and subjective appetite ratings of two different lunch meal treatments in two separate participant groups fed different protein rich meals: 1. Meat-derived protein meal, and 2. Plant-derived protein meal using a randomized, two-period, within participants, crossover design. The two test conditions for each protein meal type will be (1) salt and pepper only preparation (No Spice, NS), and (2) herb and spice preparation (Spice, S). Within each protein meal type, the two test meals will be matched for macronutrients and calories. Each participant will consume either the meat meal or the vegetarian meal at both of their two testing days that will be at least one week apart. Each participant will be randomized into a meal type sequence group so that the order of consuming the No Spice or Spice meals will be randomized.
Who Masked: Participant, Investigator
Masking Description: Test meal items will be identical except for the addition of culinary spices. Meals will be prepared by Nutrition Core Laboratory staff who have no contact with participants. Meals will be coded and given to study staff to serve to participants. Entree appearance may differ due to presence of culinary herbs (green specks) and may have different aroma. However, the PI will not be present during meal testing and thus will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meat based protein, no spice (Active Comparator): Test meal will be a chicken salad entree consisting of shredded skinless chicken breast, mayonnaise, lemon juice, celery, salt and pepper, with whole wheat crackers and grapes as side items.
  Interventions: Other: Meat based protein with added spice; Plant based protein with added spice
- Meat based protein, spice added (Experimental): Test meal will be a chicken salad entree consisting of shredded skinless chicken breast, mayonnaise, lemon juice, celery, salt and pepper, onion powder, garlic powder, dill and ground mustard seed, served with whole wheat crackers and grapes as side items.
  Interventions: Other: Meat based protein with added spice; Plant based protein with added spice
- Plant based protein, no spice (Active Comparator): Test meal will be a chick pea and rice salad entree consisting of chick peas, brown rice, mayonnaise, yogurt, lemon juice, celery, soy protein powder, salt and pepper, served with whole wheat crackers and grapes as side items.
  Interventions: Other: Meat based protein with added spice; Plant based protein with added spice
- Plant based protein, spice added (Experimental): Test meal will be a chick pea and rice salad entree consisting of chick peas, brown rice, mayonnaise, yogurt, lemon juice, celery, soy protein powder, salt and pepper, onion powder, garlic powder, cumin, parsley, dill, oregano, ground rosemary and ground mustard seed, served with whole wheat crackers and grapes as side items.
  Interventions: Other: Meat based protein with added spice; Plant based protein with added spice

INTERVENTIONS:
Other: Meat based protein with added spice; Plant based protein with added spice — Either meat or plant based protein entrees will have herbs and spices added (in addition to salt and pepper in the base recipe) to intensify the flavor profile in order to see if protein consumption is affected.

SUMMARY:
To evaluate whether or not high quality protein intake from a mixed meal can be increased by using culinary herbs and spices to increase flavor intensity and food item liking in older adults.

DETAILED DESCRIPTION:
There are two specific aims:

1. To assess whether healthy older adults ≥60 years are able to consume 1.2g/kg/BW of high quality protein (the suggested requirement for older adults) in a single meal (lunch, accounting for approximately 30% of total daily energy intake).
2. To assess whether protein intake at a single meal is increased by enhancing the flavor intensity and perceived liking of the protein rich food using culinary herbs and spices.

The hypothesis is that it is feasible to meet the suggested increased protein requirement for older adults of 1.2 g/kg/BW (Baum et al.) (at 30% of daily energy/meal) in a single meal and that addition of culinary spices results in greater perceived flavor intensity and liking and greater intake compared to a meal prepared with only salt and pepper.

ELIGIBILITY:
Inclusion criteria:

* Adults ≥ 60 years
* All body weights
* Regularly consume lunch ≥5 d/wk

Exclusion Criteria:

* Diagnosed taste or sensory disorders that would prevent evaluating the food
* Known eating disorders
* Allergies to the test food/ingredients (including herbs and spices)
* Medications or medical conditions that may adversely affect taste (e.g., dysgeusia)
* Inability to complete the protocol
* Dietary restrictions re. test meal items/ingredients (e.g., prescribed low salt diet)
* Dislike of the particular food items or herb/spices to be served in the test meals

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Protein consumption at lunch test meal | 45 minute test lunch meal on either visit one or visit two (spice or no spice in random order)
  Grams of protein consumed per kg body weight at lunch test meal. Grams of protein consumption will be determined from the amount of each food item consumed multiplied by the protein density (g protein per gram food item) of each item. Amount consumed will be determined by subtracting the weight of any food item not consumed from the weight of each food item provided. Protein density will be determined by calculating the grams of protein 100 grams of food item using ingredient information for the entree and the U. Minnesota Nutrition Data System (NDS) tables for protein content of ingredients, NDS tables for grapes and using manufacturer's information for the whole wheat crackers. Body weights will be measured at the beginning of visit one to the testing center using a calibrated body weight scale.

SECONDARY OUTCOMES:
Subjective liking of protein entree and entire meal | At completion of 45 minute lunch test meal on visits one and two (spice or no spice in randomized order)
  Participants will fill out a two item check list using a 9-point hedonic scale rating the liking of the entree item and of the entire meal The scale is a 9-point likert scale with scores ranging from 1 - 9 to assess liking (where the lowest rating of 1 indicated extreme disliking and the highest rating of 9 indicated extreme liking).
Subjective appetite ratings following lunch test meal | At completion of 45 minute lunch test meal on visits one and two (spice or no spice in randomized order)
  Participants will complete a four item visual analog scale (VAS) asking about hunger, fullness, desire to eat and prospective consumption. Each item will consist of a 100mm horizontal scale anchored at each end by "not at all hungry" and "extremely hungry"; "not at all full" and "extremely full"; "no desire to eat" and "extreme desire to eat"; and "not much at all" and "an extreme amount".
Subjective rating of flavor intensity of lunch entree and overall meal | At completion of 45 minute lunch test meal on visits one and two (spice or no spice in randomized order)
  Participants will complete a two item check list using a 5 point Likert scale rating the flavor intensity of the entree and overall meal. The scale will be anchored at one end by "no intensity at all" and at the other by "extremely intense".

CONTACTS AND LOCATIONS:
Overall Officials: John C Peters, PhD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- Anschutz Health and Wellness Center Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baum JI, Kim IY, Wolfe RR. Protein Consumption and the Elderly: What Is the Optimal Level of Intake? Nutrients. 2016 Jun 8;8(6):359. doi: 10.3390/nu8060359. PMID 27338461